CLINICAL TRIAL: NCT04337645
Title: Resective Surgical Treatment of Peri-implantitis. A Randomized Controlled Clinical Trial.
Brief Title: Resective Surgical Treatment of Peri-implantitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Belgrade (Other)
Collaborators: George Eastman Dental Hospital, Italy (Other)
Responsible Party: Principal Investigator, Iva Milinkovic, Assisstant Professor, University of Belgrade
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22101980
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Two treatment modalities will be applied. Test group will be treated bu resective approach combined with implantoplastry, whilst control group will be treated by resective approach alone. Randomization will be performed by means of randomisation envelopes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): resective surgical treatment of peri-implantitis (decontamination performed with titanium brushes and sterile saline) combined with implantoplasty
  Interventions: Procedure: surgical treatment of peri-implantitis
- Control group (Active Comparator): resective surgical treatment of peri-implantitis (decontamination performed with titanium brushes and sterile saline)
  Interventions: Procedure: surgical treatment of peri-implantitis

INTERVENTIONS:
Procedure: surgical treatment of peri-implantitis — resective surgical treatment of peri-implantitis

SUMMARY:
Surgical treatment of peri-implantitis can be regenerative or resective, depending on defect configuration. The aim of resective therapy of peri-implantitis is to reduce the severity of soft tissue inflammation and stabilize crestal bone levels whilst reducing probing depths.This will be a multicenter randomized controlled trial in which two resective peri-implantitis protocols will be assessed. The aim of this trial is to compare a resective approach in the surgical treatment of peri-implantitis (decontamination performed with titanium brushes and sterile saline) with a resective approach combined with implantoplasty.

DETAILED DESCRIPTION:
The aim of the present multicenter randomized controlled trial is to compare a resective approach in the surgical treatment of peri-implantitis (decontamination performed with titanium brushes and sterile saline) with a resective approach combined with implantoplasty.

Primary outcome:

Probing depth (PD) dicrease is defined as the primary pitcome of this study.

Research Hypothesis Based upon previous evidence, our research hypothesis is that the test group (implantoplasty + resective approach) will perform better than the control group (resective surgery alone), namely the alternative hypothesis, in terms of defect resolution (probing depth decrease, absence of bleeding and/or suppuration and absence of progressive bone loss), 18 months after the surgical treatment.

Material and methods The present study has a prospective, multicenter, randomized controlled clinical trial design in which subjects will be consecutively enrolled according to defined inclusion and exclusion criteria. Two centers participating in this study are: Department of Periodontics and Oral Medicine, School of Dental Medicine, University of Belgrade and Department of Periodontology and Protshodontics, Eastman Dental Hospital, Policlinico Umberto I, Rome, Italy.

28 patients diagnosed with severe peri-implantitis and requiring surgical treatment of peri-implantitis will be included in this study.

14 patients with peri-implantitis will be treated in each center. The subjects willing to participate in the study will be given a detailed description of the procedure and follow-up appointments, and will sign a written informed consent form. CONSORT (Consolidated Standards of Reporting Trials) guidelines for clinical trials will be followed.

Treatment groups

The patients will be randomly divided into two groups:

* Test group: resective surgery with bone recontouring + implantoplasty
* Control group: resective surgery with bone recontouring+ decontamination protocol (Ti brush and sterile saline) The randomization- and therefore the group assignment of the patient- will be disclosed after flap reflection. The randomization sequence will be generated by a computer program.

Blinding: due to the nature of the implantoplasty procedure, it is not possible to blind the outcome assessors because the plastied surface is easily recognizable compared to a rough, non-plastied surface.

Treatment protocol:

* Consent followed by clinical examination, evaluation of inclusion and exclusion criteria.
* If the patient is included, diagnosis, radiographic and photographic documentation collection. Diagnosis will be assigned after a complete periodontal chart of all teeth and implants is performed. This will be executed once the prosthetic restoration is removed. Once the clinical visit is concluded the prosthesis will be replaced.
* Baseline examination with clinical parameters' recording. Clinical parameters will be recorded by a single examiner, different from the surgeon.
* Non-surgical treatment of peri-implantitis by means of professional cleaning of teeth and implants, scaling and root planing, and CHX mouth rinse, to decrease inflammation.
* Collection of clinical parameters and evaluation of the study defect. Initially the defect will be evaluated pre-surgically. If the surgical inspection of the defect reveals that it does not have the desired characteristics (Class II, eventually Class IIIa and Class IIIb), the defect will be treated according to a regenerative surgical protocol, (the patient will therefore be excluded from the study and exempted from all future study procedures). In alternative, if deemed hopeless the implant may also be removed.
* Removal of prosthesis and placement of healing abutments, to be kept after the surgical procedure unless the implant is visible, and it is esthetically mandatory to deliver the prosthesis.
* Surgical procedure:

Following local anesthesia application, intrasulcular incisions will be performed, and full-thickness flaps shall be reflected on the buccal and lingual aspects of the affected implants. After the exposure of the implants, thorough degranulation of the defect by means of titanium and carbon curettes will be performed, followed by sterile saline rinses.

Test group implants will be treated by means of implantoplasty. Exposed threads of the implant will be removed by the protocol proposed by Ramel et al: diamond burs (106-, 40-, 15-mm) followed by Arkansas stone. Copious sterile saline irrigation will follow. Following the implantoplasty procedure, CHX gel 0.2% will be applied for 2 minutes.

In the control group, a decontamination protocol containing mechanical debridement with Ti-brush, followed by sterile saline solution on cotton pellets and CHX gel 0.2% for 2 minutes, followed by thorough rinsing with saline will be applied.

Think about local antimicrobial application, there is a product called GelCide, we started using it here at the Department The suprabony component in both groups will be removed and bone recontouring will be performed, when indicated. Mucoperiosteal flaps will be adjusted and closed with single interrupted sutures. Prosthetic constructions will be reconnected. Patients will be prescribed systemic antibiotic (Augmentin 1 g twice per day) for 1 week and 0.2% CHX rinse, twice daily, for 14 d following surgery. If the patient is allergic to penicillins, clindamycin 300 mg TID will be used instead). The duration of the surgery (time in minutes) will also be recorded.

Clinical measurements:

At baseline, as well as 6, and 12, and 18 months following the surgical treatment, following data will be acquired:

1. Clinical attachment level (CAL), distance in millimeters from:

   In the case of bone-level implants implant-abutment connection to the deepest probing point (mm). In the case of tissue level implants, CAL will be measured as the distance between the smooth-rough surface interface to the deepest probing point (mm)
2. Probing depth (PD), measured as distance from the mucosal margin to the bottom of the probeable pocket (mm).
3. Bleeding on probing (BOP), evaluated as present if bleeding was evident within 30 s after probing, or absent, if no bleeding was noticed with- in 30 s after probing. Profuse bleeding will be recorded based upon recent evidence that many implant have pinpoint bleeding even if healthy, which could possibly be due to tissue trauma.
4. Plaque index by Silness and Loe.
5. Mucosal recession on buccal aspect of the implant; bone level implants: distance from the implant platform to the gingival margin; Tissue level implants: distance between the smooth-rough surface interface to the gingival margin (mm).
6. Keratinized tissue width (KTW), as the distance from mucosal margin to the mucogingival line at the buccal and lingual aspect of each implant, 4 sites per implant (mm).
7. Keratinized tissue thickness (KTT). This will be measured clinically, with an endodontic file with silicon disc stop and a digital caliper. The measurement will be conducted in the mesial line angle (m), distal line angle (d) and mid-buccal (b), in mm.

Radiographic analysis: radiographs will be conducted at baseline/ pre-surgical, 6 months, 12 months, 18 months, 24 months. Intraoral radiographs will be performed with a standardized technique to ensure that the periapicals are comparable for each patient between consecutive time-points.

Photographic documentation: photographs will be conducted at baseline/ pre-surgical, 3 months, 6 months, 12 months, 18 months, 24 months.

Expected outcomes - Success criteria The resolution of peri-implant disease, treatment success, will be defined as probing pocket depth ≤5 mm, absence of bleeding and/or suppuration on probing, and no additional bone loss (when comparing the 2 week radiograph and the 6-, 12- and 18-month radiograph).

The success criteria proposed by Buser et al. and Cochran et al. will be followed as well at each recall after the treatment. An implant will be considered successful if shows:

i. absence of clinically detectable mobility ii. absence of pain or any other subjective sensation iii. absence of recurrent peri-implant infection iv. absence of continuous peri-implant radiolucency.

ELIGIBILITY:
Inclusion Criteria:

* · Patients >18 years old, able to provide consent and willing to undergo study procedures.

  * Implants in function for at least 1 year.
  * Patients with implant-supported partial/full jaw restorations having at least one implant diagnosed with peri-implantitis (probing pocket depth [PPD] ≥6mm, bleeding/suppuration on probing [BoP/SoP+] and marginal bone loss >2 mm compared to a previous radiographic examination or marginal bone level >3 mm (Berglundh et al. 2018)
  * Patients with suprabony defects and intrabony defects up to 3mm in depth
  * Retrievability of prosthetic reconstructions prior the surgical treatment (i.e. screw-retained restorations or cement-retained restorations which can easily be removed prior to all study visits)
  * According to classification by Monje (Monje, 2019), implants presenting Class II, eventually Class IIIa and Class IIIb
  * No implant mobility
  * No evidence of occlusal overload
  * Satisfactory oral hygiene level (FMPS<25%) and periodontal health or localized periodontal inflammation (FMBS<30%)
  * Treated periodontal disease with adequate periodontal supportive therapy

Exclusion Criteria:

* · Patients unable or unwilling to comply with study procedures and study visits.

  * Pregnant or nursing women
  * Local conditions that may interfere with surgical treatment (non-treated periodontal disease, acute infections, carious lesions, etc.)
  * Compromised systemic health preventing the patient from attending study visits or representing a contraindication for surgical treatment
  * Patients with uncontrolled systemic conditions which may affect healing (i.e. diabetes mellitus). Diabetic patients will have to document their level of metabolic control by means of HbA1c and will only be included when HbA1c<7%.
  * Patients smoking more than 5 cigarettes per day (self-reported)
  * Patients taking medications known to interfere with gingival or bone metabolism (e.g. calcium channel blockers, bisphosphonates).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
probing depth | 18 months
  measured distance in milimeters from the mucosal margin to the bottom of the probeable pocket (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Iva Milinkovic, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code